CLINICAL TRIAL: NCT06557044
Title: The Analgesic Efficacy of Pericapsular Nerve Group (PENG) Block in Patients Undergoing Primary Total Hip Arthoplasty: a Prospective, Double-blinded, Randomized Controlled Trial
Brief Title: The Analgesic Efficacy of Pericapsular Nerve Group (PENG) Block in Patients Undergoing Primary Total Hip Arthoplasty:
Acronym: PENG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Diakonie-Klinikum Stuttgart (Other)
Collaborators: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Prof. Dr. Rainer Meierhernich, Principal Investigator, Diakonie-Klinikum Stuttgart
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Diak 001/2024
Record Dates: First submitted 2024-08-08; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Prospective; Randomized; Double-blind
Keywords: Pericapsular Nerve Group Block; hip endoprostheses
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum Group (Experimental): 20 ml ropivacaine 0.5%
  Interventions: Drug: Ropivacaine
- Placebo Group (Placebo Comparator): 20 ml physiological saline
  Interventions: Other: Physiological saline

INTERVENTIONS:
Drug: Ropivacaine — PENG block with ropivacaine
  Arms: Verum Group
Other: Physiological saline — Placebo control
  Arms: Placebo Group

SUMMARY:
The aim of this study is to investigate the analgesic efficacy of the pericapsular nerve group (PENG) block during the implantation of hip endoprostheses. The study is designed as a prospective randomized double-blind study and the study participants were randomized into 2 arms and either 20 ml ropivacaine 0.5% (verum group) or 20 ml physiological saline solution (placebo group) will be applied.

ELIGIBILITY:
Inclusion Criteria:

* planned cementless hip TEP operation for primary coxarthrosis via minimally invasive anterolateral approach using the identical implant system (Taperloc stem, Plamafit cup)
* Patient capable of giving consent
* Informed consent has been obtained
* age > 18 years

Exclusion Criteria:

* Refusal to participate in the study
* Regular use of opioids
* Known chronic pain symptoms
* Infections in the area of the puncture site
* Presence of a contraindication to ropivacaine
* Presence of a contraindication to metamizole
* Presence of a contraindication to postoperative analgesia with diclofenac
* Secondary forms of osteoarthritis with deformities (i.e. high-grade dysplasia, secondary conditions after trauma, secondary conditions after childtrauma, secondary conditions after childhood hip joint diseases
* Spinopelvic dysbalance, spinal canal stenosis
* Previous operations on the hip/pelvis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Rate of postoperative opioid administration | 60 minutes after arrival in the recovery room
  The primary objective is to investigate the influence of the PENG block on the need for postoperative ntravenously opioid administration within the first hour in the recovery room.

SECONDARY OUTCOMES:
Quantity of total opioid consumption | until the evening of the second postoperative day
  Assessment of total opioid consumption until second postoperative day in both arms
Intensity of postoperative pain | until the evening of the second postoperative day
  Subjective perception of postoperative pain, using the numeric rating scale.
Intensity of postoperative nausea and vomiting | until the evening of the second postoperative day
  Assessment of postoperative nausea/vomiting using the PONV Score
Postoperative recovery | until the evening of the second postoperative day
  Assessment of postoperative recovery using the QoR15 score

CONTACTS AND LOCATIONS:
Locations (1):
- Diakonie-Klinikum Stuttgart, Stuttgart, Baden-Wurttemberg, Germany